CLINICAL TRIAL: NCT06957652
Title: Reconstructive Treatment of Combined Peri-implantitis-related Defects With or Without Collagen Membrane: A Randomized Clinical Study
Brief Title: Reconstructive Treatment of Peri-implantitis With Combined Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sıla Çağrı İşler, Associate Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-KAEK-27/04
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Peri-implantitis
Keywords: Reconstructive therapy; peri-implantitis; Bone defect; barrier membrane
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Active Comparator): Reconstructive surgical therapy of combined peri-implantitis defects using a resorbable collagen membrane and DBMM-C.
  Interventions: Device: DBMM-C plus Resorbable collagen membrane
- Control group (Active Comparator): Reconstructive surgical therapy of combined peri-implantitis defects using only DBMM-C.
  Interventions: Device: DBMM-C

INTERVENTIONS:
Device: DBMM-C plus Resorbable collagen membrane — A trapezoidal flap design will be employed, including a sulcular incision and vertical releasing incisions extending approximately 2-3 mm beyond the mucogingival junction. Flap advancement will be facilitated through a periosteal-releasing incision at the flap base. Granulation tissue will be removed using a titanium curette, and implant surface decontamination will be performed with a titanium brush. The graft material will be placed in both supra- and intrabony defect components, followed by coverage with a resorbable collagen membrane. The flaps will then be coronally advanced and stabilized over the biomaterials.
  Arms: Test Group
Device: DBMM-C — A trapezoidal flap design will be employed, including a sulcular incision and vertical releasing incisions extending approximately 2-3 mm beyond the mucogingival junction. Flap advancement will be facilitated through a periosteal-releasing incision at the flap base. Granulation tissue will be removed using a titanium curette, and implant surface decontamination will be performed with a titanium brush. The graft material will be placed in both supra- and intrabony defect components, and then the flaps will be coronally advanced and stabilized over the graft material.
  Arms: Control group

SUMMARY:
The aim of this randomized clinical study is to assess the additional clinical benefit of incorporating a resorbable collagen membrane (CM) alongside a xenogeneic bone graft-specifically, deproteinized bovine bone mineral with 10% collagen (DBBM-C)-in the reconstructive surgical treatment of peri-implantitis involving combined (i.e., contained and non-contained) defect configurations.

Accordingly, the study addresses the following research questions:

* Does the adjunctive use of a CM in combination with DBBM-C improve treatment success compared to DBBM-C alone in the management of combined peri-implantitis-related defects?
* Does the combined use of a CM and DBBM-C lead to superior patient-reported outcomes (PROs) compared to the use of DBBM-C alone in the reconstructive treatment of such defects? A total of 60 patients who have been referred to the Gazi University Department of Periodontology will be randomly assigned to receive test (DBMM-C +CM) or control group (DBMM-C) treatments. Clinical parameters will be assessed at baseline (i.e., prior to surgery), and at the 6-, and 12-month post-operatively. Radiographic examinations will be carried out at baseline and 12 months post-operatively. Patient oral health related to the treatment procedures will be evaluated using a written questionnaire [Oral Health Impact Profile (OHIP-14)] prior to treatment and after 2 weeks, 1, and 12 months following surgical therapy. Regarding post-treatment pain and overall patient satisfaction with treatment modalities, responses will be scored on a visual analog scale (VAS, 100 mm).

DETAILED DESCRIPTION:
Reconstructive surgical therapy for peri-implantitis has shown improved clinical and radiographic outcomes, with favorable postoperative mucosal margin levels and superior radiographic bone fill compared to other treatment modalities. However, no specific biomaterial or application technique has yet been identified as clearly superior. In particular, the potential added value of combining a barrier membrane with a bone substitute, as opposed to using bone substitute alone, remains a subject of ongoing debate.

Recent studies have suggested that the adjunctive use of a barrier membrane does not necessarily enhance clinical or radiographic outcomes in peri-implantitis-associated intrabony defects. However, these studies often included heterogeneous defect morphologies, which may influence the regenerative potential and confound treatment outcomes.

Indeed, "contained" and "non-contained" defects may behave differently due to biological factors such as space maintenance, clot stability, and wound protection. his highlights the need to tailor biomaterial selection to the specific defect configuration. While current evidence suggests that barrier membranes may not provide additional benefit in fully contained defects, there is a lack of data regarding their effectiveness in combined defects that include both supracrestal and intrabony components, particularly those with partially contained 2- or 3-wall morphologies.

Therefore, the primary aim of this randomized clinical study is to evaluate the additional clinical benefit of incorporating a resorbable CM with DBMM-C in the reconstructive surgical treatment of peri-implantitis with combined defect morphology.

The secondary objective is to assess patient-reported outcomes (PROs) in both treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Peri-implantitis defined as the presence of a peri-implant probing pocket depth (PPD) ≥6 mm with bleeding and/or suppuration on probing (BoP/SoP) and radiographic marginal bone loss (MBL) ≥3 mm.
* Presence of combined defect configuration Class [Ib, Ic, Ie with horizontal components (i.e. Class II) (Schwarz et al., 2010)] with an intrabony compartment of ≥3 mm.
* Presence of a minimum width of 2 mm of keratinized peri-implant mucosa on the buccal aspect of the implant.
* Implants placed in proper position (inside the bony housing)
* Having an implant-supported prosthesis that allows for adequate oral hygiene procedures and peri-implant probing.

Exclusion Criteria:

* Full-mouth plaque score (FMPS) < 25%
* Full-mouth bleeding score (FMBS) < 25%
* Cigarette smoking < 10 cig./day,
* Diagnosed with active periodontal disease,
* Having acute or chronic medical conditions or undergoing medications, such as intravenous amino-bisphosphonates, immunosuppressive drugs, and chemotherapy, that could interfere with the treatment outcome,
* Receiving antibiotic treatment in the previous 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of treatment success (%) | 12 months after the surgical treatment
  The absence of bleeding on probing (BOP) at more than one site, no suppuration, deepest PPD ≤5mm, and no further radiographic bone loss.

SECONDARY OUTCOMES:
Percentage of bleeding on probing (BOP) (%) | 12 months after the surgical treatment
  The percentage of BOP around six sites of the implant
Probing pocket depth (PPD) | 12 months after the surgical treatment
  The distance between the bottom of the pocket and the mucosal margin around the implant
Change in radiographic vertical defect depth | 12 months after the surgical treatment
  Marginal bone levels (MBL) will be assessed the distance between this line and the first bone-to-implant contact (BIC). The mesial and distal measurements will be averaged for further calculations. The radiographic vertical defect depth changes over time will be evaluated the difference between MBL at baseline and 12 months following the therapy.
Patient morbidity - Postoperative pain | At baseline and after 2 weeks and 1 and 12 months following surgical treatment
  Postoperative pain will be assessed using a visual analogue score
Patient-reported satisfaction with the overall treatment | At baseline and after 2 weeks and 1 and 12 months following surgical treatment
  Patient-reported satisfaction will be assessed using a visual analogue score

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Dentistry, Ankara, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Regidor E, Ortiz-Vigon A, Romandini M, Dionigi C, Derks J, Sanz M. The adjunctive effect of a resorbable membrane to a xenogeneic bone replacement graft in the reconstructive surgical therapy of peri-implantitis: A randomized clinical trial. J Clin Periodontol. 2023 Jun;50(6):765-783. doi: 10.1111/jcpe.13796. Epub 2023 Mar 6. PMID 36802084
- [Background] Schwarz F, Becker K, Albrecht C, Ramanauskaite A, Begic A, Obreja K. Effectiveness of modified and control protocols for the surgical therapy of combined peri-implantitis-related defects. A retrospective analysis. Clin Oral Implants Res. 2023 May;34(5):512-520. doi: 10.1111/clr.14057. Epub 2023 Mar 10. PMID 36852537
- [Background] Raabe C, Cafferata EA, Couso-Queiruga E, Chappuis V, Ramanauskaite A, Schwarz F. Impact of Two Flap Advancement Techniques and Periosteal Suturing on Graft Displacement During Guided Bone Regeneration. Clin Implant Dent Relat Res. 2025 Feb;27(1):e13434. doi: 10.1111/cid.13434. PMID 39815673